CLINICAL TRIAL: NCT02876900
Title: A Randomized, Double-Blind, Placebo-Controlled, Fixed-Dose, 6-Week, In-Patient Study to Assess Efficacy and Safety of HP-3070 in Subjects Diagnosed With Schizophrenia
Brief Title: Study to Assess Efficacy and Safety of HP3070 in Subjects Diagnosed With Schizophrenia.
Acronym: HP-3070
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Noven Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Noven Therapeutics (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HP-3070-GL-04
Record Dates: First submitted 2016-08-03; First posted 2016-08-24 (Estimated); Results first posted 2020-03-27 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Transdermal Patch

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low dose Asenapine maleate patch (Experimental): Low dose asenapine maleate, transdermal patches will be compared against placebo patches.
  Interventions: Drug: Low Dose Asenapine maleate transdermal patch; Drug: Placebo
- High dose asenapine maleate patch (Experimental): High dose asenapine maleate, transdermal patches will be compared against placebo patches.
  Interventions: Drug: High Dose Asenapine maleate transdermal patch; Drug: Placebo
- Placebo transdermal patch (Placebo Comparator): Low dose or high dose asenapine maleate transdermal patch will be compared against placebo patches
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Low Dose Asenapine maleate transdermal patch — The study will evaluate low dose Asenapine maleate transdermal patch
  Other Names: Transdermal patch
  Arms: Low dose Asenapine maleate patch
Drug: High Dose Asenapine maleate transdermal patch — The study will evaluate high dose Asenapine maleate transdermal patch
  Other Names: Transdermal patch
  Arms: High dose asenapine maleate patch
Drug: Placebo — The study will evaluate placebo transdermal patch.
  Other Names: Sham treatment

SUMMARY:
This study is designed to evaluate efficacy and safety of HP-3070 compared with placebo transdermal patch in subjects diagnosed with schizophrenia.

DETAILED DESCRIPTION:
This is a Phase 3, randomized, double-blind, placebo-controlled, in-patient, efficacy, and safety study to evaluate HP-3070 for the treatment of schizophrenia.

This study is designed to evaluate efficacy and safety of HP-3070 compared with placebo transdermal patch in subjects diagnosed with schizophrenia, who are in an acute exacerbation and to assess the impacts of covariates on asenapine exposure as delivered in a patch formulation, using a population-based approach.

ELIGIBILITY:
Inclusion Criteria:

* Current diagnosis of schizophrenia.
* Subject has PANSS total score ≥80, AND score of 4 or more in at least 2 of the following PANSS items at Screening and at Baseline: conceptual disorganization delusions; hallucinatory behavior; unusual thought content.
* Subjects must be able to wear a transdermal patch for 24 hours.

Exclusion Criteria:

* Subject has been diagnosed with schizophrenia less than 6 months prior to Screening Visit.
* Subject has received within 90 days of Screening Visit: electroconvulsive therapy; transcranial magnetic stimulation; vagal nerve stimulation; or other brain stimulation treatments
* Subject has experienced acute depressive symptoms within 30 days prior to Screening Visit that requires treatment with an antidepressant, as determined by the Investigator.
* Currently taking clozapine for the treatment of schizophrenia.
* Has hypothyroidism or hyperthyroidism.
* Subject is currently being treated with insulin for diabetes.
* Subject has epilepsy or history of seizures.
* Positive urine pregnancy test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 617 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Harb, MD, MPH, Study Director — Noven Pharmaceuticals, Inc.
Locations (1):
- Noven Pharmaceuticals, Inc., Jersey City, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Citrome L, Komaroff M, Starling B, Byreddy S, Terahara T, Hasebe M. Efficacy of HP-3070, an Asenapine Transdermal System, on Symptoms of Hostility in Adults With Schizophrenia: A Post Hoc Analysis of a 6-Week Phase 3 Study. J Clin Psychiatry. 2022 Jun 6;83(4):21m14355. doi: 10.4088/JCP.21m14355. PMID 35687858
- [Derived] Citrome L, Walling DP, Zeni CM, Starling BR, Terahara T, Kuriki M, Park AS, Komaroff M. Efficacy and Safety of HP-3070, an Asenapine Transdermal System, in Patients With Schizophrenia: A Phase 3, Randomized, Placebo-Controlled Study. J Clin Psychiatry. 2020 Dec 15;82(1):20m13602. doi: 10.4088/JCP.20m13602. PMID 33326711

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Dose Asenapine Maleate Patch: Low dose asenapine maleate, transdermal patches will be compared against placebo patches.
  Low Dose Asenapine maleate transdermal patch: The study will evaluate low dose Asenapine maleate transdermal patch.
  Placebo: Evaluate Low Dose versus Placebo.
- High Dose Asenapine Maleate Patch: High dose asenapine maleate, transdermal patches will be compared against placebo patches.
  High Dose Asenapine maleate transdermal patch: The study will evaluate high dose Asenapine maleate transdermal patch
  Placebo: Evaluate High Dose versus Placebo.
- Placebo Patch: Placebo transdermal patch
Period: Overall Study
Arm/Group | Low Dose Asenapine Maleate Patch | High Dose Asenapine Maleate Patch | Placebo Patch
Started | 205 | 206 | 206
Completed | 166 | 158 | 162
Not Completed | 39 | 48 | 44

BASELINE CHARACTERISTICS:
Population: A total of 616 subjects were randomized in the double-blind treatment period of the study and were included in the Intent-to-Treat (ITT) analysis set (206 patients in HP-3070 18.0 mg group, 204 patients in HP-3070 9.0 mg group, 206 patients in placebo group). One additional subject met exclusion criteria for the study but was not dosed (n=617).
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose Asenapine Maleate Patch | High Dose Asenapine Maleate Patch | Placebo Patch | Total
Number analyzed (Participants) | 204 | 206 | 206 | 616
Age, Customized [Count of Participants; unit: Participants]
  <55 | 168 | 172 | 171 | 511
  >=55 | 36 | 34 | 35 | 105
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 95 | 75 | 243
  Male | 131 | 111 | 131 | 373
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 5 | 1 | 16
  Not Hispanic or Latino | 194 | 201 | 205 | 600
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: A total of 616 subjects were randomized in the study and were included in the ITT analysis set. For Race, a subject could select more than one race in the case report form.
  Participants
    American Indian or Alaska Native | 0 | 1 | 0 | 1
    Asian | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 47 | 45 | 54 | 146
    White | 157 | 159 | 152 | 468
    More than one race | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 61 | 62 | 62 | 185
  Russia | 60 | 60 | 60 | 180
  Bulgaria | 29 | 30 | 29 | 88
  Ukraine | 35 | 35 | 36 | 106
  Serbia | 19 | 19 | 19 | 57
Height [Mean (Standard Deviation); unit: cm] | 172.5 (9.08) | 171.8 (9.09) | 171.8 (9.16) | 172.0 (9.10)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 26.591 (5.1151) | 26.240 (4.7834) | 25.925 (4.8602) | 26.251 (4.9205)
PANSS total score [Count of Participants; unit: Participants] — Population: Safety Analysis Set = 614 subj who received double-blind medication. PANSS total score is sum of all 30 items (7 positive items, 7 negative items & 16 general psychopathology items). For each item, severity rated on an anchored 7-point scale; score of 1=absence of symptoms, score of 7=extremely severe symptoms. Total score ranges from 30 to 210.
  Participants
    number analyzed (Participants) | 204 | 204 | 206 | 614
    <90 | 45 | 53 | 54 | 152
    >=90 | 159 | 151 | 152 | 462

OUTCOME MEASURES:

1. Primary Outcome: Evaluate Efficacy and Safety of Asenapine Maleate Patches Compared With Placebo Patches in Subjects Diagnosed With Schizophrenia as Measured Using the Syndrome Scale (PANSS) Total Score: Change From Baseline to Week 6.
Description: To evaluate efficacy and safety of HP-3070 compared with placebo for the treatment of schizophrenia as evaluated by Positive and Negative Syndrome Scale (PANSS) total score.
  The PANSS total score is the sum of all 30 items (7 positive items, 7 negative items, and 16 general psychopathology items). For each item, severity was rated on an anchored 7-point scale, with a score of 1 indicating the absence of symptoms and a score of 7 indicating extremely severe symptoms. If one or more items are missing at a given assessment, the total score is set to missing. Total score ranges from 30 to 210. Score indicates severity of the disease, i.e. low score = low severity.
Time Frame: 6 weeks
Population: Results are from the full analysis set (FAS) which includes all randomized participants who had at least 1 patch of double-blind study medication applied and who have a baseline PANSS total score and at least 1 post baseline assessment of the primary efficacy measure (PANSS total score) and completed the study.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Low Dose Asenapine Maleate Patch | High Dose Asenapine Maleate Patch | Placebo Patch
Number analyzed (Participants) | 201 | 203 | 203
score on a scale | -22.1 (1.158) | -20.4 (1.162) | -15.5 (1.166)
Statistical Analysis 1: Comparison: High Dose Asenapine Maleate Patch vs Placebo Patch; The mixed model for repeated measures includes treatment, country, visit, treatment by visit interaction, and baseline value as covariates, and participant as random effect. The correlation of repeated measures within a participant is estimated with an unstructured covariance matrix. The Kenward-Rogers method is used to estimate the denominator degrees of freedom; Test type: Superiority — Assuming an effect size of 0.35 on the change in PANSS total score from baseline to Week 6 for the 2 pairwise comparisons between each active asenapine maleate transdermal patch treatment arm and placebo, the power for detecting a statistically significant HP-3070 advantage was approximately 0.90, having 204 evaluable participants per each treatment arm using a 2-sided alpha level of 0.025 for each comparison; p = 0.003, Mixed Model Repeated Measures Analysis — Adjusted p-value was calculated according to the truncated Hochberg procedure with a truncation factor y=0.9. Adjustment for multiple comparisons uses a parallel gatekeeping procedure; Least Square Mean Difference = -4.8, 95% CI 2-sided [-8.06 to -1.64], Standard Error of Mean 1.634
Statistical Analysis 2: Comparison: Low Dose Asenapine Maleate Patch vs Placebo Patch; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 1, analysis 1]; Least Square Mean Difference = -6.6, 95% CI 2-sided [-9.81 to -3.4], Standard Error of Mean 1.63

2. Secondary Outcome: Evaluate Efficacy and Safety of Asenapine Maleate Patches Compared With Placebo Patches in Subjects Diagnosed With Schizophrenia as Measured Using the Clinical Global Impression - Severity of Illness Scale: Change From Baseline to Week 6.
Description: To evaluate efficacy and safety of HP-3070 compared with placebo for the treatment of schizophrenia as evaluated by the Clinical Global Impression - Severity of Illness Scale.
  The severity of illness for each participant was rated using the CGI-S. The rater or Investigator answered the following question: "Considering your total clinical experience with this particular population, how mentally ill is the participant at this time?". Response choices included: 0 = not assessed; 1 = normal, not at all ill, 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; and 7 = among the most extremely ill participants.
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Dose Asenapine Maleate Patch | High Dose Asenapine Maleate Patch | Placebo Patch
Number analyzed (Participants) | 201 | 203 | 203
score on a scale | -1.3 (0.90) | -1.2 (0.96) | -0.9 (0.93)
Statistical Analysis 1: Comparison: High Dose Asenapine Maleate Patch vs Placebo Patch; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Mixed Model Repeated Measures Analysis — Adjusted p-value was calculated according to the Hochberg procedure. Adjustment for multiple comparisons uses a parallel gatekeeping procedure; Least Square Mean Difference = -0.4, 95% CI 2-sided [-0.55 to -0.16], Standard Error of Mean 0.1
Statistical Analysis 2: Comparison: Low Dose Asenapine Maleate Patch vs Placebo Patch; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Least Square Mean Difference = -0.4, 95% CI 2-sided [-0.64 to -0.25], Standard Error of Mean 0.099

ADVERSE EVENTS:
Time Frame: From date of first dose of doubleblind (DB) study medication (Day 1) through the 30 day follow-up period, approximately 72 days.
Description: The safety analysis set included all participants who had at least 1 patch of double-blind study medication applied and who have at least 1 post dose safety measurement during the double-blind treatment period.
Groups:
- Placebo: Placebo transdermal patch
Arm/Group | Low Dose Asenapine Maleate Patch | High Dose Asenapine Maleate Patch | Placebo
All-Cause Mortality (participants affected / at risk) | 0/204 | 0/204 | 0/206
Serious Adverse Events (participants affected / at risk) | 3/204 | 2/204 | 4/206
Other Adverse Events (participants affected / at risk) | 75/204 | 78/204 | 70/206
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose Asenapine Maleate Patch (N=204) | High Dose Asenapine Maleate Patch (N=204) | Placebo (N=206)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Acute Coronary Syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal ulcer hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Schizophrenia (Psychiatric disorders) | 2 (2) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose Asenapine Maleate Patch (N=204) | High Dose Asenapine Maleate Patch (N=204) | Placebo (N=206)
Weight increased (Investigations) | 8 (8) | 12 (12) | 4 (4)
Headache (Nervous system disorders) | 18 (23) | 19 (21) | 13 (13)
Extrapyramidal disorder (Nervous system disorders) | 13 (16) | 19 (22) | 3 (4)
Application site erythema (General disorders) | 19 (105) | 20 (57) | 3 (14)
Constipation (Gastrointestinal disorders) | 11 (12) | 9 (11) | 9 (10)
Insomnia (Psychiatric disorders) | 15 (21) | 14 (16) | 23 (28)
Anxiety (Psychiatric disorders) | 10 (14) | 11 (13) | 13 (19)
Agitation (Psychiatric disorders) | 5 (5) | 6 (7) | 11 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-01-20): https://cdn.clinicaltrials.gov/large-docs/00/NCT02876900/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-18): https://cdn.clinicaltrials.gov/large-docs/00/NCT02876900/SAP_001.pdf